CLINICAL TRIAL: NCT00229593
Title: A Randomized, Open Label Clinical Trial to Evaluate if Nestorone Gel Has Gonadotropin Suppressive Activity and if Nestorone in Combination With Testosterone Will Have an Additive Effect on Gonadotropin Suppression When Applied Transdermally in Healthy Men
Brief Title: NES Gel-1, To Evaluate Nestorone Gel in Combination With Testosterone Gel
Acronym: NES-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, William Bremner, Study Principal Investigator, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 26852-D; HHSN27500002;; 04-3792-D 02 (Other: UW Human Subjects Division)
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Contraception
Keywords: Male contraception; Androgen; Progestin; Spermatogenesis; Gonadotropin suppression; Testosterone; Nestorone
MeSH Terms: interventions — Testosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- 1 (Active Comparator): 100 mg Testosterone gel daily for 3 weeks
  Interventions: Drug: Testosterone Gel
- 2 (Active Comparator): 2 mg Nestorone gel daily for 3 weeks
  Interventions: Drug: Nestorone gel
- 3 (Active Comparator): 4 mg Nestorone gel daily for 3 weeks
  Interventions: Drug: Nestorone gel
- 4 (Active Comparator): 100 mg Testosterone gel + 2 mg Nestorone gel
  Interventions: Drug: Nestorone gel; Drug: Testosterone Gel
- 5 (Active Comparator): 100 mg Testosterone gel + 4 mg Nestorone gel
  Interventions: Drug: Nestorone gel; Drug: Testosterone Gel
- 6 (Active Comparator): 100 mg Testosterone Gel + 6 mg Nestorone Gel daily for 3 weeks
  Interventions: Drug: Nestorone gel; Drug: Testosterone Gel
- 7 (Active Comparator): 100 mg Testosterone Gel + 8 mg Nestorone gel daily for 3 weeks
  Interventions: Drug: Nestorone gel; Drug: Testosterone Gel

INTERVENTIONS:
Drug: Nestorone gel — 2 to 8 mg Nestorone gel daily for 3 weeks depending on treatment group assignment
  Arms: 2; 3; 4; 5; 6; 7
Drug: Testosterone Gel — 100 mg Testosterone gel daily for 3 weeks
  Other Names: Testim
  Arms: 1; 4; 5; 6; 7

SUMMARY:
The purpose of this study is to determine the usefulness of two transdermal gels to be used in the future development for a male contraceptive.

DETAILED DESCRIPTION:
The success of hormonal male contraception depends on the near complete suppression of spermatogenesis without producing any untoward effects on libido or other androgen-dependent functions or any other adverse events. The treatment with androgen alone has geen shown to be highly effective in Asian men but less effective in non-Asian men in clinical trials. To increase the efficacy of androgen alone treatment on spermatogenesis, combined regimens of a progestin and an androgen have shown promising results. The steady-state delivery of a progestin and an androgen by transdermal gel application would be a user-friendly delivery method as compared to injectable or implant approaches. Nestorone (NES) is a synthetic progestin that does not have any androgenic and estrogenic activity and is not expected to have some of the undesirable side effects of other drugs.

We propose to evaluate whether NES gel alone or in combination with T gel applied transdermally will result in more effective suppression of gonadotropins than NES or T gel applied alone in healthy men. Fifty healthy male subjects, age 18-50 will be enrolled at each center (2 sites).

ELIGIBILITY:
Inclusion Criteria:

* Healthy men
* Aged 18-50 years
* With normal clinical chemistry, serum levels of testosterone, PSA, gonadotropins within normal limits, and sperm concentration greater than 20 million/mL
* Subject or his partner willing to use a recognized effective method of contraception

Exclusion Criteria:

* Men not living in area of clinics
* Clinically significant abnormal findings at screening
* Elevated PSA greater than 4
* Partners who are pregnant
* Abnormal laboratory values, liver or kidney dysfunction
* Sperm counts below 20 million/mL.
* Use of androgens or body building substances within 6 months of enrollment,
* Blood pressure greater than 140/90, history of hypertension, including hypertension controlled with treatment
* History of primary testicular disease or disorder of the hypothalamic-pituitary axis
* Hypersensitivity of progestins
* History of venous thromboembolism
* Benign or malignant liver tumors
* Active liver disease, history of reproductive dysfunction including vasectomy or infertility
* History of active or chronic cardiac, renal, hepatic or prostatic disease
* Diabetes mellitus or morbid obesity (body weight greater than 120% of ideal body weight)
* Known or suspected alcoholism or drug abuse
* Known dermatitis or severe skin disorder

Men desiring fertility within 6 months or participating in competitive sports where drug screening for prohibited substances (including anabolic steroids) is routine will be advised of the relative and temporary hazards that participating in this study may have for their fertility or sporting status.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2005-09; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
- To determine the gonadotropin suppressive activity of Nestorone (NES) Gel at two doses and T gel at one dose alone or in combination over a 3-week period. Serum levels of gonadotropins will be assessed in all subjects. | 3 weeks

SECONDARY OUTCOMES:
To determine the effects on serum levels of total and free testosterone and SHBG and measure serum levels of NES gel. | 3 weeks
Safety measured laboratory evaluations, vitals, pre- and post treatment physical exam results and PSA levels | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: William J Bremner, MD, PhD, Principal Investigator — University of Washington; Christina Wang, MD, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - Harbor-UCLA Medical Center, Torrance, California
  - University of Washington Medical Center, Seattle, Washington

REFERENCES:
- [Background] Anawalt BD, Bebb RA, Bremner WJ, Matsumoto AM. A lower dosage levonorgestrel and testosterone combination effectively suppresses spermatogenesis and circulating gonadotropin levels with fewer metabolic effects than higher dosage combinations. J Androl. 1999 May-Jun;20(3):407-14. PMID 10386821
- [Background] Anderson RA, Kinniburgh D, Baird DT. Suppression of spermatogenesis by etonogestrel implants with depot testosterone: potential for long-acting male contraception. J Clin Endocrinol Metab. 2002 Aug;87(8):3640-9. doi: 10.1210/jcem.87.8.8773. PMID 12161488
- [Background] Bebb RA, Anawalt BD, Christensen RB, Paulsen CA, Bremner WJ, Matsumoto AM. Combined administration of levonorgestrel and testosterone induces more rapid and effective suppression of spermatogenesis than testosterone alone: a promising male contraceptive approach. J Clin Endocrinol Metab. 1996 Feb;81(2):757-62. doi: 10.1210/jcem.81.2.8636300.
- [Background] Brache V, Massai R, Mishell DR, Moo-Young AJ, Alvarez F, Salvatierra AM, Cochon L, Croxatto H, Robbins A, Faundes A. Ovarian function during use of Nestorone(R) subdermal implants. Contraception. 2000 Mar;61(3):199-204. doi: 10.1016/s0010-7824(00)00092-5. PMID 10827334
- [Background] Cummings DE, Bremner WJ. Prospects for new hormonal male contraceptives. Endocrinol Metab Clin North Am. 1994 Dec;23(4):893-922. PMID 7705326
- [Background] Diaz S, Schiappacasse V, Pavez M, Zepeda A, Moo-Young AJ, Brandeis A, Lahteenmaki P, Croxatto HB. Clinical trial with Nestorone subdermal contraceptive implants. Contraception. 1995 Jan;51(1):33-8. doi: 10.1016/0010-7824(94)00006-i. PMID 7750282
- [Background] Gonzalo IT, Swerdloff RS, Nelson AL, Clevenger B, Garcia R, Berman N, Wang C. Levonorgestrel implants (Norplant II) for male contraception clinical trials: combination with transdermal and injectable testosterone. J Clin Endocrinol Metab. 2002 Aug;87(8):3562-72. doi: 10.1210/jcem.87.8.8710. PMID 12161475
- [Background] Haukkamaa M, Laurikka-Routti M, Heikinheimo O, Moo-Young A. Contraception with subdermal implants releasing the progestin ST-1435: a dose-finding study. Contraception. 1992 Jan;45(1):49-55. doi: 10.1016/0010-7824(92)90140-o. PMID 1591921
- [Background] Handelsman DJ, Conway AJ, Howe CJ, Turner L, Mackey MA. Establishing the minimum effective dose and additive effects of depot progestin in suppression of human spermatogenesis by a testosterone depot. J Clin Endocrinol Metab. 1996 Nov;81(11):4113-21. doi: 10.1210/jcem.81.11.8923869.
- [Background] Kamischke A, Heuermann T, Kruger K, von Eckardstein S, Schellschmidt I, Rubig A, Nieschlag E. An effective hormonal male contraceptive using testosterone undecanoate with oral or injectable norethisterone preparations. J Clin Endocrinol Metab. 2002 Feb;87(2):530-9. doi: 10.1210/jcem.87.2.8218. PMID 11836281
- [Background] Kamischke A, Venherm S, Ploger D, von Eckardstein S, Nieschlag E. Intramuscular testosterone undecanoate and norethisterone enanthate in a clinical trial for male contraception. J Clin Endocrinol Metab. 2001 Jan;86(1):303-9. doi: 10.1210/jcem.86.1.7057. PMID 11232016
- [Result] Mahabadi V, Amory JK, Swerdloff RS, Bremner WJ, Page ST, Sitruk-Ware R, Christensen PD, Kumar N, Tsong YY, Blithe D, Wang C. Combined transdermal testosterone gel and the progestin nestorone suppresses serum gonadotropins in men. J Clin Endocrinol Metab. 2009 Jul;94(7):2313-20. doi: 10.1210/jc.2008-2604. Epub 2009 Apr 14. PMID 19366848